CLINICAL TRIAL: NCT06629467
Title: Cognitive Behavioral Treatment with Activity Trackers for Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Alba González-Roz, PhD, Professor, PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SV-PA-21-AYUD/2021/50884.
Record Dates: First submitted 2024-07-29; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use Cessation; Physical Activity
Keywords: Tobacco; Physical activity; Activity tracker; Cognitive-behavioral therapy
MeSH Terms: conditions — Tobacco Use Cessation; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1) CBT for smoking cessation + personalized PA plan + Fitbit Versa 3 ®. (Experimental): The intervention will be delivered in groups (maximum 4 participants) for a total of 6 weeks. Sessions (1.5 hours) will take place once per week. Personalized PA objectives will be set during the treatment.
  Participants in this arm will wear the Fitbit Versa 3® during the treatment (6 weeks).
  Interventions: Behavioral: Cognitive-behavioral therapy for smoking cessation; Behavioral: Personalized PA plan; Device: Fitbit Versa 3
- 2) CBT for smoking cessation + personalized PA plan (Active Comparator): This intervention include the same components as described above. The exception will be that participants will not be requested to wear the Fitbit Versa 3®.
  Interventions: Behavioral: Cognitive-behavioral therapy for smoking cessation; Behavioral: Personalized PA plan

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy for smoking cessation — Treatment components will include psychoeducation on the consequences of tobacco use and the benefits of quitting; therapeutic commitment; self-monitoring of cigarette smoking; brief advice on healthy eating behaviors and sleep hygiene, physiological feedback (based on CO levels), training in self-control strategies, stimulus control, management of craving with alternative activities, diaphragmatic breathing, weekly personalized physical activity objectives, and relapse prevention strategies. The protocol consists of a nicotine fading procedure, which consists of a weekly reduction in nicotine intake of 30% (based on both tobacco brands and the number of cigarettes) from the first to the fifth session.
Behavioral: Personalized PA plan — The treatment provider will fix an objective (e.g. go for brisk walking for 30 minutes 3 times this week) for each participant every week according to his/her current PA level, time availability, likes, and fitness level.
Device: Fitbit Versa 3 — Wearable activity tracker with the functionalities of a watch function, including time, date, calendar, and weather (connection to the internet is required). Physical activity monitoring (steps per day, active minutes per day, plants climbed, heart rate monitoring, time, intensity, caloric expenditure, and exercise type of exercise session), sleep monitoring (sleep time, sleep phases time, sleep quality), stress levels managing and guided breathing application are the main health-related functionalities.
  Arms: 1) CBT for smoking cessation + personalized PA plan + Fitbit Versa 3 ®.

SUMMARY:
Given the high prevalence of deaths per year attributable to tobacco use, improving smoking cessation treatments is an important public health priority Worldwide. It is also known that practicing physical activity (PA) may help smoking cessation. Physical activity trackers have been demonstrated to increase PA levels in different studies with various populations, as a sole intervention or in combination with interventions targeting PA.

This study aims to examine the feasibility, effect, and cost-effectiveness of cognitive-behavioral therapy (CBT) + Personalized physical activity (PA) + Physical Activity Tracker use (Fitbit Versa 3®) for smoking cessation. Given the high prevalence of deaths per year attributable to tobacco use, improving smoking cessation treatments is an important public health priority worldwide.

In this study, an estimated sample of 128 adult smokers will be randomly allocated to one of the following conditions: 1) CBT for smoking cessation + personalized PA plan + Fitbit Versa 3®; 2) CBT for smoking cessation + personalized PA plan.

Mail goals: 1) To examine the feasibility (i.e., adherence, perceived utility, satisfaction) of integrating Fitbit Versa 3® into a CBT protocol for smoking cessation; 2) to examine the effectiveness of CBT for smoking cessation + personalized PA plan + Fitbit Versa 3® and CBT for smoking cessation + personalized PA plan in terms of smoking abstinence rates (point-prevalence and days of continuous abstinence), PA (i.e., steps per day, moderate to vigorous physical activity) and mental health outcomes (anxiety and depression symptoms, emotional dysregulation); 3) to examine the cost-effectiveness of CBT for smoking cessation + personalized PA plan + Fitbit Versa 3® vs. CBT for smoking cessation + personalized PA plan in terms of smoking abstinence rates (point-prevalence and days of continuous abstinence), PA (i.e., steps per day, moderate to vigorous physical activity) and mental health outcomes (anxiety and depression symptoms, emotional dysregulation).

DETAILED DESCRIPTION:
Fitbit® wearables devices inform on several objective data related to physical activity and sleep habits, amongst others. Incipient research has piloted its use for vulnerable populations such as emerging adults and clinical patients. In the field of substance use, some studies looked at the effects of activity trackers on physical activity but did not evaluate its effects on other clinically relevant variables, such as smoking abstinence. Increases in activity and improvements in mood are associated with smoking abstinence and, arguably, using Fitbit Versa 3® devices would produce any effect on cigarette smoking via these variables.

A 6-week protocol will be employed including a cognitive behavioral therapy-based smoking cessation treatment. Participants will be recruited from the community and will be randomly allocated to the following conditions once an in-person assessment is completed: 1) CBT for smoking cessation + personalized PA plan + Fitbit Versa 3®; 2) CBT for smoking cessation + personalized PA plan. According to the power analysis, to detect an effect size of d = 0.5 (medium size effect) with a test power of 0.8 the total number of allocated participants will be 128. This sample size was estimated to be sufficient for the statistical pipeline.

Analyses will be conducted using the Statistical Package for the Social Science (SPSS), R Studio, JASP, and JAMOVI. A set of univariate (i.e., descriptive statistics and frequencies) and multivariate analyses (i.e. t-test) will be carried out with regard to participants; characteristics and treatment outcomes. Generalized Estimating Equations (GEE) will be conducted to examine changes in smoking abstinence after controlling for relevant covariates (e.g., nicotine dependence, sex). DATCAP will be used to perform the cost-effectivity

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 or over.
* Smoking at least 10 cigarettes per day.

Exclusion Criteria:

* Being currently receiving other psychological or pharmacological treatment for smoking cessation.
* Being diagnosed with substance use disorder or severe psychiatric disorder.
* Active suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the activity tracker | End-of-treatment (6-weeks)
  Acceptability of the activity tracker is measured using the Participant Experience Questionnaire (PEQ) at the end of treatment. This scale ranges from 10 to 50. A higher score means higher acceptability.
Tobacco use | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  This variable is operationalized as changes in cigarettes/day, carbon monoxide (CO) changes, and self-reported and verified abstinence (i.e., ≤4 ppm).
Feasibility of treatment and activity tracker use | End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Feasibility is operationalized as treatment completion, attendance to sessions and adherence to Fitbit Versa 3 use.
Physical activity | In-treatment, from enrollment to end-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Physical activity (PA) is operationalized as steps per day, plants climbed per day, distance covered per day (kilometers), light physical activity (minutes per day), moderate physical activity (minutes per week), vigorous physical activity (minutes per week), and sedentary time (hours per day). These outcomes will be measured using an adapted version of the International Physical Activity Questionnaire (IPAQ) and Fitbit Versa 3®.
Activity tracker perceived utility | End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Perceived utility with the activity tracker is measured using dichotomous (yes/no) ad-hoc; questions about the utility of the activity tracker for smoking cessation, increasing physical activity, and improving sleep quality.

SECONDARY OUTCOMES:
Anxiety symptoms | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Anxiety symptoms are measured using Generalized Anxiety Disorder-7 (GAD-7). This questionnaire ranges from 0 to 21. Higher punctuation means higher anxiety levels symptoms.
Depression symptoms | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Depression symptoms are measured using the Patient Health Questionnaire-9 (PHQ-9). This questionnaire ranges from 0 to 14. A higher punctuation means higher depression symptom levels.
Hypothetical demand for cigarettes | Enrollment
  CPT (Cigarette purchase task) (Items: Maximum number of cigarettes smoked per day, maximum expenditure in cigarettes per day and maximum expenditure per pack)
Emotional dysregulation of negative valence emotions | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Emotional dysregulation of negative emotions is measured with the Difficulties in emotion regulation scale-16 (DERS-16). This scale ranges from 16 to 80 points. A higher score means more difficulties in emotion regulation of negative valence emotions.
Emotional dysregulation of positive valence emotions | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Emotional dysregulation of positive emotions is measured with Difficulties in Emotion Regulation Scale-Positive (DERS-P). This scale ranges from 13 to 65. A higher score means more difficulties in emotion regulation of positive valence emotions.
Delay Discounting | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  Single and cross-commodity computerized Delay Discounting task of money and tobacco (delay of one day, one week, one month and six month time)
Suicide ideation | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  This variable is measured with the Paykel suicide ideation scale (PSS). This scale ranges from 0 to 5 points. Higher punctuation means more severe suicide ideation.
Life Quality | From Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  This variable is measured with the European quality of life- 5 dimensions- 5 levels (EQ-5D-5L). This scale ranges from 5 to 25. A higher score means less life quality (more health-related problems).
Sleep quality | In treatment (6 weeks), from Enrollment to End-of-treatment (6-weeks), one-, three-, six-, -month follow-up.
  This variable is measured using The Pittsburgh Sleep Quality Index (PSQI). This scale ranges from 0 to 21 points. A higher score means lower sleep quality. In addition, Fitbit Versa 3 provides a sleep quality punctuation ranging from 0 to 100. A higher punctuation means better sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Unit of Addictive Behaviors, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Abrantes AM, Van Noppen D, Bailey G, Uebelacker LA, Buman M, Stein MD. A Feasibility Study of a Peer-Facilitated Physical Activity Intervention in Methadone Maintenance. Ment Health Phys Act. 2021 Oct;21:100419. doi: 10.1016/j.mhpa.2021.100419. Epub 2021 Aug 14. PMID 34552664
- [Background] Carreiro S, Chintha KK, Shrestha S, Chapman B, Smelson D, Indic P. Wearable sensor-based detection of stress and craving in patients during treatment for substance use disorder: A mixed methods pilot study. Drug Alcohol Depend. 2020 Apr 1;209:107929. doi: 10.1016/j.drugalcdep.2020.107929. Epub 2020 Mar 3. PMID 32193048
- [Background] Goldfine C, Lai JT, Lucey E, Newcomb M, Carreiro S. Wearable and Wireless mHealth Technologies for Substance Use Disorder. Curr Addict Rep. 2020 Sep;7(3):291-300. doi: 10.1007/s40429-020-00318-8. Epub 2020 Jun 11. PMID 33738178
- [Background] Purani H, Friedrichsen S, Allen AM. Sleep quality in cigarette smokers: Associations with smoking-related outcomes and exercise. Addict Behav. 2019 Mar;90:71-76. doi: 10.1016/j.addbeh.2018.10.023. Epub 2018 Oct 17. PMID 30368021